CLINICAL TRIAL: NCT03348215
Title: The Design and Testing of a Targeted, Treadmill Based Training Program for Post-Stroke Gait Rehabilitation, Through Co-Production With Users; Incorporating Visual Flow, and Functional Electrical Stimulation
Brief Title: Enhanced Treadmill Gait Training With Lower Limb Support After Stroke
Acronym: ENTRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Strathclyde (Other)
Responsible Party: Principal Investigator, Andrew Kerr, Principal Investigator, University of Strathclyde
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SU_BME_KERR01102017
Record Dates: First submitted 2017-10-02; First posted 2017-11-20 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: Gait rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This is a singles subject design with participants acting as their own control. Control data being recorded during the week before the intervention begins
Masking Description: The primary gait measure (number of daily steps in teh community) will be collected by an independent assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced Treadmill Training (Other): Treadmill walking with an immersive environment and bio mechanical support (body weight, ankle-foot -orthosis and functional electrical stimulation)
  Interventions: Other: Enhanced Treadmill Training

INTERVENTIONS:
Other: Enhanced Treadmill Training — 6 week programme of treadmill training with addition of an immersive environment (virtual reality projection), body weight support, orthotics and functional electrical stimulation

SUMMARY:
This series of single case studies aims to test the feasibility and acceptability of an enhanced treadmill system for the recovery of gait function in stroke survivors. Forty adult participants who have had a stroke in the past year that resulted in impaired gait function and are attending a local hospital for gait training, will be recruited. Participants will be asked to attend a rehabilitation clinic for seven weeks, three times a week where they will receive enhanced treadmill training supervised by a physiotherapist. Assessment sessions will take place in week 1, weeks 5 and 8, and after 3 months. Outcome measures recorded during assessment sessions will include gait variables (e.g. speed, cadence, step length and joint kinematics) measured overground and on the treadmill using motion capture technology and outside using body worn sensors (inertial motion unit). Participants will complete a questionnaire on their community walking habits and asked to wear a physical activity monitor for 48 hours to record stepping time.

The basic intervention will comprise of walking on a treadmill capable of adjusting its speed to match that of the user (using feedback from the motion capture system) and a large television screen showing a virtual reality scene (woodland walking) with visual perturbations (virtual obstacle avoidance). In addition participants will be divided equally and randomly (Latin square) to either wear an ankle foot orthosis (AFO group) or functional electrical stimulation (FES group) while walking on the treadmill but not provided for home use. Training sessions will last up to a max of 20 minutes, will be supervised by a physiotherapist and participants will wear a safety harness to remove any risk of trip falls. Any adverse event such as muscle/joint pain, illness or a fall at home will be recorded, participants and physiotherapists will also be asked for feedback on their experience with the treadmill system using questionnaires and semi-structured interviews

DETAILED DESCRIPTION:
Design Series of single case studies investigating feasibility and acceptability of an enhanced treadmill training system incorporating self pacing, virtual reality and biomechanical support with either an ankle foot orthosis (AFO) or functional electrical stimulation (FES) which will be decided using a Latin square.

Participants Individuals referred to rehabilitation services due to impaired walking function resulting from a stroke in the past 12 months and who are medically stable, will be invited to participate.

Target sample size = 40. Eligible participants will be approached about participation by a clinical trials nurse who will allow at least 48 hours for consideration before giving consent. The percentage of eligible people invited to participate who then agree to participate will be noted as the recruitment rate.

Outcome measures Following informed consent, participants will be asked to attend a physiotherapy gym at a local hospital for a total of eight consecutive weeks, three times a week with a follow assessment 3 months later.

Outcome measures will be recorded at weeks 1, 5, 8 and 20. These will include:

1. Physical activity recorded over 48 hours using an accelerometer based sensor worn on the thigh (ActivPal, PalTechnologies, Glasgow, UK).
2. Spatiotemporal gait variables (walking speed, cadence, step length, stride length, stance duration) during treadmill, overground indoor and overground outdoor walking using a combination of motion capture technology (Vicon, Oxford Metrics, Oxford, UK) and inertial sensors (Trigno, Delsys, Mass, USA).
3. Lower limb 3D joint angles during treadmill, overground indoor and overground outdoor walking using a combination of motion capture technology (Vicon, Oxford Metrics, Oxford, UK) and inertial sensors (Trigno, Delsys, Mass, USA).
4. Acceptability of the intervention using bespoke satisfaction questionnaires and semi structured interviews with the therapists and participants.
5. Adverse and serious adverse events such as falls, illness, joint/muscle soreness will be recorded as part of the routine research governance but also to assess acceptability and feasibility.
6. Community walking ability using a standard questionnaire (Perry, J., et al. (1995). "Classification of Walking Handicap in the Stroke Population," Stroke 26(6): 982-989.) and a semi structured interview.

Intervention The core of the intervention will be walking on a self-pacing, single belt, treadmill (N-mill, Motekforce link, Amsterdam) in front of a large (65 inch) high definition screen (Dell, USA) which will show a virtual reality scene (woodland walk) synchronised with the belt speed to provide an immersive walking environment. The treadmill is surrounded by six motion capture cameras (VICON, Oxford Metrics, Oxford, UK) which capture the three dimensional movement of markers placed on the lower limbs and trunk of the individual. These data are used to control the belt speed and provide performance feedback to therapists/patients either in real time through visualisation on the screen or afterwards when the data are fully processed. Using a Latin square to remove selection bias participants will be further allocated to either receive an ankle foot orthosis (AFO group) or functional electrical stimulation (FES group), both of which will be used only during the treadmill. training. At the initial assessment visit participants will be examined for skin damage or impaired circulation in the lower leg and foot which would exclude them from using an AFO or FES.

FES group A dual-channel surface electrical stimulator (NeuroTrac® Rehab, Model number: ECS305A) will be used to stimulate four major muscle groups; the ankle dorsiflexors and plantarflexors, and the knee flexors and extensors. The FES will be triggered using real time data from the motion capture system. The physiotherapist will decide which muscle groups should be used to support gait training and the timing and amplitude of the FES administered. Participants will be excluded from the FES group if they have any implants in the vicinity of the FES sites. These participants will be transferred to the AFO group if they are agreeable. Skin integrity will be check at each treatment visit before and after the intervention. Should signs of skin trauma present the intervention will discontinued and the participant provided with advice and referred to their general practitioner if considered appropriate by the physiotherapists.

AFO group A standard AFO (polypropylene posterior leaf) will be fitted under the guidance of the physiotherapist and orthotist. A range of sizes (small, medium, large and extra ) will be available (Complete care shop, Lancashire, UK) which will be adjusted using heel raises so that the lower leg has an angle of 10-12 degrees to the vertical at the point of mid stance. The AFO will be worn during the treadmill walking only. If participants are already using an AFO they will continue to use this as before.

Duration Duration will be determined by the supervising physiotherapist based on the participant's tolerance. The aim will be to increase incrementally to a maximum of 20 minutes of continuous walking.

Frequency Frequency will be determined by the supervising physiotherapist based on tolerance of the participant and practical issues such as transport. The aim will be to attend three times a week.

The treadmill training (AFO and FES groups) will replace any conventional gait training provided by the therapists, however, any unrelated training e.g. Upper limb exercises or speech therapy will continue as normal practice.

Intensity Walking speed will be set at a comfortable pace. Initially this will be 80% of their overground indoor walking assessed at week one. Speed will be increased incrementally as appropriate and advised by the physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old.
2. Have had a diagnosed stroke.
3. Onset of stroke between 1 week and 12 months prior to recruitment.
4. Attending Coathill Hospital (NHS Lanarkshire) for stroke rehabilitation which includes gait training.
5. Have Hemiplegia.
6. Medically Stable.
7. Able to follow simple, verbal instructions in English, or in another language if an appropriate translator is available.
8. Able to provide informed consent.

Exclusion Criteria:

1. Considered by the GP or NHS clinicians to be unsafe to do mild exercise for the duration of time required (about 20 minutes).
2. Have contracture of the hip, knee or ankle which prevents walking.
3. Have any skin irritation on the shank.
4. Have a cardiac pacemaker.
5. A body mass that exceeds the capacity of the equipment (>100Kg).
6. Cognitive impairment severe enough to prevent adherence with the protocol (assessed by the clinicians responsible for each volunteer).
7. Walking difficulty before stroke (for example, patients who had history of severe spinal stenosis or peripheral vascular diseases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Participant compliance with the intervention | 12 months
  Proportion of participants attending 60% of training sessions.

SECONDARY OUTCOMES:
Community walking ability | 12 months
  The Walking Ability Questionnaire:
  This questionnaire measures ability to walk in the community/home. (Perry et al (1995). Stroke, 26(6), pp.982-989.) This is a questionnaire based on self reported ability in 19 ambulatory activities , 8 in the home and 11 in the community. Each activity has an associated ordinal scale of ability ranging from "unable" to "independent". The overall score ranges between 0 and 76 with higher scores equating to better community walking.
Physical activity behaviour | 12 months
  Time spent lying, sitting, standing and walking during a 48 hour period using an established physical activity monitor (ActivPal, PalTechnologies, Glasgow, Scotland)
Gait performance | 12 months
  Speed, step length, cadence, lower limb angles. Measured by motion capture system (Vicon, Oxford, UK) indoors (overground and treadmill) and outdoors with body mounted sensors (Trigno, Delsys, Mass. USA)
Participant satisfaction with the enhanced treadmill training. | 12 months
  Satisfaction questionnaires using 5 point ordinal scales of satisfaction. 7 Items related to the intervention, such as the virtual reality projection, are rated on an ordinal scale. An overall score between 0 and 25 is calculated with a higher score indicating greater satisfaction.
Participants satisfaction with the intervention and overall research experience | 12 months
  Semi structured interviews:
  Participant's opinions will be sought regarding the intervention and their overall experience in this research study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kerr, PhD, Principal Investigator — University of Strathclyde
Locations (1):
- Coathill Hospital, Coatbridge, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phongamwong C, Rowe P, Chase K, Kerr A, Millar L. Treadmill training augmented with real-time visualisation feedback and function electrical stimulation for gait rehabilitation after stroke: a feasibility study. BMC Biomed Eng. 2019 Aug 22;1:20. doi: 10.1186/s42490-019-0020-1. eCollection 2019. PMID 32903355